CLINICAL TRIAL: NCT07170969
Title: A Feasibility Trial of an Enhanced Coping-oriented Supportive Programme (E-COSP) for Community-Dwelling People With Spinal Cord Injury
Brief Title: A Feasibility Trial of an Enhanced Coping-oriented Supportive Programme for Community-dwelling People With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PolyuSNLIYAN
Record Dates: First submitted 2025-09-04; First posted 2025-09-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury; Mental Health; Feasibility Studies; Acceptability Study; Spinal Cord Injuries (SCI); Spinal Cord Injuries; Coping
Keywords: spinal cord injuries; feasibility and acceptability; mental health; Participation in meaningful activities; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We aim to have a single study group, which the group will receive eight weekly online group sessions (6-8 participants per group) with one hour for each session using Zoom videoconferencing software.
Masking Description: There is only one study group, and the trial will estimate the feasibility and acceptability of the E-COSP during the pre and post intervention. Therefore, all participants and investigators not necessary to be blinded due to the nature of this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Feasibility Trial of an Enhanced Coping-oriented Supportive Programme (E-COSP) for Community-Dwell (Experimental): The E-COSP intervention, modified from the original COSP, consists of eight weekly online group sessions via Zoom. Its four components-orientation, cognitive appraisal, coping strategies (4 sessions), and social support (2 sessions)-are enhanced with realistic community scenarios and strengthened self-efficacy training. A trained rehab nurse with over three years of SCI experience will deliver the manualized intervention. The nurse will receive extensive training and ongoing supervision from experts and a psychologist. Intervention fidelity will be ensured through audio-taped session reviews by the principal investigators.
  Interventions: Other: An Enhanced Coping-oriented Supportive Programme (E-COSP) for Community-Dwelling People with Spinal Cord Injury

INTERVENTIONS:
Other: An Enhanced Coping-oriented Supportive Programme (E-COSP) for Community-Dwelling People with Spinal Cord Injury — The intervention group will receive eight weekly online group sessions (6-8 participants per group) with one hour for each session using Zoom videoconferencing software. A detailed intervention manual will be used to guide all intervention delivery. The intervention will be led by a registered rehabilitation nurse (who will be employed as a part-time RA2) who has more than three years of work experience in caring for people with SCI. The nurse who delivers the intervention will receive extensive training from the PI and CI, who are experts in coping interventions and relevant psychosocial intervention skills. The intervention providers will also receive training in group dynamics and group intervention skills, and be supervised by the research team and a psychologist during the whole period of the study. Selected audio-taped intervention sessions will be rated by the PI and CI on the fidelity of the intervention delivery

SUMMARY:
Spinal cord injury (SCI) is a neurological disorder that leads to "partial or complete loss of people's motor and/ or sensory function below the level of the injury".

This study is a single-group feasibility trial with pre- and post-assessment. The total sample size is 12. This is a feasibility trial of an Enhanced Coping-oriented Supportive Programme (E-COSP) for Community-Dwelling People with Spinal Cord Injury.

Twelve SCI participants will be recruited from the Hong Kong Direction Association for the Handicapped. The intervention group will receive eight weekly online group sessions (6-8 participants per group) with one hour for each session using Zoom videoconferencing software. A detailed intervention manual will be used to guide all intervention delivery. The intervention will be led by a registered rehabilitation nurse (who will be employed as a part-time RA2) who has more than three years of work experience in caring for people with SCI. The nurse who delivers the intervention will receive extensive training from the PI and CI, who are experts in coping interventions and relevant psychosocial intervention skills. The intervention providers will also receive training in group dynamics and group intervention skills, and be supervised by the research team and a psychologist during the whole period of the study. Selected audio-taped intervention sessions will be rated by the PI and CI on the fidelity of the intervention delivery.

Primary outcome will be the feasibility and acceptability: The feasibility will be assessed by recruitment rate, retention rate, and drop-out rate; and the acceptability will be assessed by adherence rate and participants' satisfaction. And the secondary outcomes will be mental health, Quality of Life, participation in meaningful activities, coping strategies, and self-efficacy.

DETAILED DESCRIPTION:
This study is a single-group feasibility trial with pre- and post-assessment. The total sample size is 12. This is a feasibility trial of an Enhanced Coping-oriented Supportive Programme (E-COSP) for Community-Dwelling People with Spinal Cord Injury.

Twelve SCI participants will be recruited from the Hong Kong Direction Association for the Handicapped. The intervention group will receive eight weekly online group sessions (6-8 participants per group) with one hour for each session using Zoom videoconferencing software. A detailed intervention manual will be used to guide all intervention delivery. The intervention will be led by a registered rehabilitation nurse (who will be employed as a part-time RA2) who has more than three years of work experience in caring for people with SCI. The nurse who delivers the intervention will receive extensive training from the PI and CI, who are experts in coping interventions and relevant psychosocial intervention skills. The intervention providers will also receive training in group dynamics and group intervention skills, and be supervised by the research team and a psychologist during the whole period of the study. Selected audio-taped intervention sessions will be rated by the PI and CI on the fidelity of the intervention delivery.

The intervention group: The E-COSP intervention includes four major components: (1) orientation and encouragement (one session); (2) cognitive appraisal (one session); (3) coping strategies (four sessions); and (4) social support and future (two sessions). The E-COSP intervention was modified from the original COSP programme. The modifications include 1) Incorporating common stressful situations or scenarios that participants may encounter in community or home settings (e.g., overcoming transportation barriers, managing social relationships with family and friends, and enhancing social participation; 2) strengthening the training content to further enhance participants' self-efficacy (e.g., effective goal setting, positive self-talk, and practical advice for skills development).

Delivery of the E-COSP intervention. The intervention group will receive eight weekly online group sessions (6-8 participants per group) with one hour for each session using Zoom videoconferencing software. A detailed intervention manual will be used to guide all intervention delivery. The intervention will be led by a registered rehabilitation nurse (who will be employed as a part-time RA2) who has more than three years of work experience in caring for people with SCI. The nurse who delivers the intervention will receive extensive training from the PI and CI, who are experts in coping interventions and relevant psychosocial intervention skills. The intervention providers will also receive training in group dynamics and group intervention skills, and be supervised by the research team and a psychologist during the whole period of the study. Selected audio-taped intervention sessions will be rated by the PI and CI on the fidelity of the intervention delivery.

Primary outcomes: Feasibility and acceptability: The feasibility will be assessed by recruitment rate, retention rate, drop-out rate; and the acceptability will be assessed by adherence rate and participants' satisfaction.

Secondary outcomes Mental health. The 14-item Hospital Anxiety and Depression Scale (HADS) will be used to assess the mental health (depression and anxiety) of the participants. The HADS comprises two subscales (each with 7 items) to assess participants' depression and anxiety levels. Responses will be given on a 0 to 3 Likert scale. Higher scores indicate more distress. Scores between 8-15 are considered mild to moderate cases, and 16 or above are severe cases. Both the Chinese and English versions of HADS have demonstrated good psychometric properties (Cronbach's alpha = 0.72-0.82) among the spinal cord injury population.

Participation in meaningful activities. The Chinese version of the Meaningful Activity Participation Assessment will be adopted. This is a checklist survey with two subscales: Frequency Subscale measures how often each activity was engaged in over the past few months on a scale from 0 (not at all) to 6 (every day); Meaningfulness Subscale assesses the perceived meaningfulness of each activity on a scale from 0 (not at all meaningful) to 4 (extremely meaningful). Scores for each item are calculated by multiplying the frequency and meaningfulness ratings, resulting in a total score ranging from 0 to 672, where higher scores indicate greater meaningful activity participation. The scale has demonstrated good psychometric properties (Cronbach's alpha = 0.86). Quality of life. The EuroQoL 5 Dimension will be adopted. This scale includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels, from no problems to extreme problems. The scale has been used in the SCI population, and it has demonstrated good psychometric properties among people with physical disabilities (Cronbach's alpha = 0.78). Coping strategies. The 28-item Coping Orientation to Problems Experienced Inventory will be used to evaluate coping strategies. This scale measures two conceptually distinct patterns of coping behaviours: maladaptive coping and adaptive coping. The score of each item ranged from 1 ('I usually do not do this at all') to 4 ('I usually do this often'). Higher scores indicated the more frequent use of the corresponding strategy. The Chinese version of this scale has demonstrated good psychometric properties (Cronbach's alpha = 0.85). Self-efficacy. The Chinese version of the Moorong Self-Efficacy Scale will be used to measure self-efficacy. It employs a seven-point Likert scale including 16 items, and the score of each item ranges from 1 to 7, with 1 indicating "very uncertain" and 7 indicating "very certain". The total score ranged from 16 to 112, with a higher score indicating more self-efficacy. This scale has demonstrated good validity among Chinese patients with SCI (Cronbach's α = 0.89).

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 -65 years old
* individuals currently living in the community with a diagnosis of SCI for at least 6 months, and who are currently having stable medical conditions
* experiencing mild to moderate depression or anxiety (scores of between 8-15 as assessed by the Hospital Anxiety and Depression Score for either the Depression or Anxiety Subscales)
* able to access and use an internet-enabled device (e.g., computer, tablet, smartphone) for attending online meetings
* able to speak/understand Cantonese/Traditional Chinese.

Exclusion Criteria:

* currently receiving any psychosocial interventions (e.g., coping skills training, cognitive behavioral therapy, or mindfulness training)
* present with any significant cognitive impairment (with reference to the clinical record), brain injury, or medical instability (with unstable cardiopulmonary diseases, pressure ulcers, contracture or marked muscle hypertonicity)
* have problems with hearing, verbal communication, and vision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the programme | Feasibility will be assessed during the post-intervention, an average of 8 weeks.
  The feasibility of the programme will be assessed by recruitment rate, retention rate, and drop-out rate.
Acceptability of the programme | Acceptability will be assessed during the post-intervention, an average of 8 weeks.
  The acceptability of the programme will be assessed by adherence rate and participants' satisfaction.

SECONDARY OUTCOMES:
Mental health at pre-intervention | Mental health will be assessed at pre-intervention, at the beginning of the study, before 8 weeks start.
  The 14-item Hospital Anxiety and Depression Scale (HADS) will be used to assess the mental health (depression and anxiety) of the participants. The HADS comprises two subscales (each with 7 items) to assess participants' depression and anxiety levels. Responses will be given on a 0 to 3 Likert scale. Higher scores indicate more distress. Scores between 8-15 are considered mild to moderate cases.
Mental health at post intervention | Mental health will be assessed at post-intervention, an average of 8 weeks.
  The 14-item Hospital Anxiety and Depression Scale (HADS) will be used to assess the mental health (depression and anxiety) of the participants. The HADS comprises two subscales (each with 7 items) to assess participants' depression and anxiety levels. Responses will be given on a 0 to 3 Likert scale. Higher scores indicate more distress. Scores between 8-15 are considered mild to moderate cases.
Participation in meaningful activities at pre-intervention | Participation in meaningful activities will be assessed at pre-intervention, at the beginning of the study, before 8 weeks start.
  The Chinese version of the Meaningful Activity Participation Assessment will be adopted [40]. This is a checklist survey with two subscales: Frequency Subscale measures how often each activity was engaged in over the past few months on a scale from 0 (not at all) to 6 (every day); Meaningfulness Subscale assesses the perceived meaningfulness of each activity on a scale from 0 (not at all meaningful) to 4 (extremely meaningful). Scores for each item are calculated by multiplying the frequency and meaningfulness ratings, resulting in a total score ranging from 0 to 672, where higher scores indicate greater meaningful activity participation.
Participation in meaningful activities at post-intervention | Participation in meaningful activities will be assessed at post-intervention, an average of 8 weeks.
  The Chinese version of the Meaningful Activity Participation Assessment will be adopted [40]. This is a checklist survey with two subscales: Frequency Subscale measures how often each activity was engaged in over the past few months on a scale from 0 (not at all) to 6 (every day); Meaningfulness Subscale assesses the perceived meaningfulness of each activity on a scale from 0 (not at all meaningful) to 4 (extremely meaningful). Scores for each item are calculated by multiplying the frequency and meaningfulness ratings, resulting in a total score ranging from 0 to 672, where higher scores indicate greater meaningful activity participation.
Quality of life at pre-intervention | Quality of life will be assessed at pre-intervention, at the beginning of the study, before 8 weeks start.
  The EuroQoL 5 Dimension will be adopted. This scale includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels, from no problems to extreme problems. The scale has been used in the SCI population, and it has demonstrated good psychometric properties among people with physical disabilities (Cronbach's alpha = 0.78).
Quality of life at post-intervention | Quality of life will be assessed at post-intervention, an average of 8 weeks.
  The EuroQoL 5 Dimension will be adopted. This scale includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels, from no problems to extreme problems. The scale has been used in the SCI population, and it has demonstrated good psychometric properties among people with physical disabilities (Cronbach's alpha = 0.78).
Coping strategies at pre-intervention | Coping strategies will be assessed at pre-intervention, at the beginning of the study, before 8 weeks start.
  The 28-item Coping Orientation to Problems Experienced Inventory will be used to evaluate coping strategies. This scale measures two conceptually distinct patterns of coping behaviours: maladaptive coping and adaptive coping. The score of each item ranged from 1 ('I usually do not do this at all') to 4 ('I usually do this often'). Higher scores indicated the more frequent use of the corresponding strategy.
Coping strategies at post-intervention | Coping strategies will be assessed at post-intervention, an average of 8 weeks.
  The 28-item Coping Orientation to Problems Experienced Inventory will be used to evaluate coping strategies. This scale measures two conceptually distinct patterns of coping behaviours: maladaptive coping and adaptive coping. The score of each item ranged from 1 ('I usually do not do this at all') to 4 ('I usually do this often'). Higher scores indicated the more frequent use of the corresponding strategy.
Self-efficacy at pre-intervention | Self-efficacy will be assessed at pre-intervention, at the beginning of the study, before 8 weeks start.
  The Chinese version of the Moorong Self-Efficacy Scale will be used to measure self-efficacy. It employs a seven-point Likert scale including 16 items, and the score of each item ranges from 1 to 7, with 1 indicating "very uncertain" and 7 indicating "very certain". The total score ranged from 16 to 112, with a higher score indicating more self-efficacy.
Self-efficacy at post-intervention | Self-efficacy will be assessed at post-intervention, an average of 8 weeks.
  The Chinese version of the Moorong Self-Efficacy Scale will be used to measure self-efficacy. It employs a seven-point Likert scale including 16 items, and the score of each item ranges from 1 to 7, with 1 indicating "very uncertain" and 7 indicating "very certain". The total score ranged from 16 to 112, with a higher score indicating more self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, Dr, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No